CLINICAL TRIAL: NCT07044583
Title: SAVE Trial: SAfe Opioid Use Video Education
Acronym: SAVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HCI186179
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Breast Reconstruction; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to a opioid video vs. no opioid video cohort by a block randomization scheme based on a predefined computer-generated sequence (six blocks, six numbers per block) in a 1:1 intervention: no intervention ratio.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid Video (Experimental): Patients in the opioid video cohort will watch a 3-minute education video on proper opioid use preoperatively. All patients who consent to study participation will be given the same surgical care and inpatient intraoperative and postoperative analgesic regimen regardless of cohort allocation.
  Interventions: Behavioral: Opioid Educational Video
- Regular Care (No Intervention): All patients who consent to study participation will be given the same surgical care and inpatient intraoperative and postoperative analgesic regimen regardless of cohort allocation.

INTERVENTIONS:
Behavioral: Opioid Educational Video — The video includes information on (1) how to consume appropriate over-the-counter pain medication alongside opioids for optimal pain control, (2) how prescribed opioids should be used only to treat pain related to the surgery, and (3) the proper disposal of unused opioids. The video was created through the University of Utah Office of Patient Experience. Feedback regarding the educational content was provided by surgeons, pain management physicians, and pharmacists throughout the process.
  Arms: Opioid Video

SUMMARY:
The study will assess the efficacy of a standardized postoperative patient-centered intervention designed to educate patients on the opioid epidemic, the judicious use of opioids, and the proper disposal of opioids. This trial is a single-institution, randomized controlled trial comparing total post-discharge opioid use in breast reconstruction patients who view an educational video on proper opioid use to patients who do not receive intentional education (the current standard of care).

This will be the first project to inform opioid prescribing guidelines for breast reconstruction patients based on actual opioid use data and will describe a patient-centered intervention that is easily incorporated into current postoperative workflows. Broadly, the results of the study aim to set the foundation to incorporate cost-effective educational interventions across multiple surgical specialties that require postoperative opioid prescription.

DETAILED DESCRIPTION:
Opioids are widely overprescribed and overused after surgery, contributing to the current opioid misuse crisis which affects more than 10 million Americans annually. In the breast reconstruction after mastectomy population, studies report as many as 47% of patients go on to become prolonged users of opioids.

The primary goal is to assess the efficacy of a standardized postoperative patient-centered intervention designed to educate patients on the opioid epidemic, the judicious use of opioids, and the proper disposal of opioids. The proposed study is a single-institution, randomized controlled trial comparing total post-discharge opioid use in breast reconstruction patients who view an educational video on proper opioid use to patients who do not receive intentional education (the current standard of care). This project is directly relevant to the mission of the AHRQ to "improve health care patient safety and to provide a 360-degree view of the patient." Specifically, this will be the first project to inform opioid prescribing guidelines for breast reconstruction patients based on actual opioid use data and will describe a patient-centered intervention that is easily incorporated into current postoperative workflows. Broadly, the results of the study aim to set the foundation to incorporate cost-effective educational interventions across multiple surgical specialties that require postoperative opioid prescription.

Patients will be randomized to an opioid video vs. no opioid video cohort by a block randomization scheme based on a predefined computer-generated sequence (six blocks, six numbers per block) in a 1:1 intervention: no intervention ratio. Patients in the opioid video cohort will watch a 3-minute education video on proper opioid use preoperatively. The video includes information on (1) how to consume appropriate over-the-counter pain medication alongside opioids for optimal pain control, (2) how prescribed opioids should be used only to treat pain related to the surgery, and (3) the proper disposal of unused opioids. The video was created through the University of Utah Office of Patient Experience. Feedback regarding the educational content was provided by surgeons, pain management physicians, and pharmacists throughout the process.

ELIGIBILITY:
Inclusion Criteria:

* Female patients 18 years of age or older
* Patients undergoing abdominally based autologous free flap breast reconstruction after mastectomy for breast cancer or cancer prophylaxis

Exclusion Criteria:

* Patients undergoing reoperations such as autologous breast reconstruction as a revision procedure following failed implant-based reconstruction
* Patients undergoing multiple procedures such as mastectomy and immediate reconstruction
* Patients with documented chronic opioid use prior to procedure, chronic pain condition

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Total Opioid Consumption | up to 2 weeks postoperative
  Total opioid consumption post-discharge from breast reconstruction, measured in Morphine Milligram Equivalents (MMEs).
Days to Opioid Cessation | up to 2 weeks postoperative
  Total number of days until ceasing opioid use from breast reconstruction surgery to 2 weeks.

SECONDARY OUTCOMES:
Opioids Prescribed Consumed | up to 2 weeks postoperative
  This outcome measure will report the percentage of opioids prescribed consumed from breast reconstruction surgery up to 2 weeks.
Non-Opioid Analgesics Consumed | up to 2 weeks postoperative
  This outcome measure will report the amount and type of non-opioid analgesics consumed from breast reconstruction surgery to 2 weeks.
Days to Non-Opioid Analgesics Cessation | up to 2 weeks postoperative
  Total number of days until ceasing of non-opioid analgesics from breast reconstruction surgery to 2 weeks.
Patient-reported Daily Pain Scores | up to 2 weeks postoperative
  Patient-reported daily pain scores from breast reconstruction surgery to 2 weeks.
  Pain Scores are numerical ratings of self-reported pain intensity from 0-10. Lower scores indicate less pain, and higher score indicate more pain.
  This outcome measure will report the mean Patient-reported Daily Pain Scores.
Complication Types | up to 2 weeks postoperative
  This outcome measure will report the frequency of the following breast reconstruction complications:
  * Poor wound healing: skin necrosis, dehiscence of wound
  * Seroma/ Hematoma
  * Infection
  * Takeback to the operating room pre-discharge
  * Unplanned readmission
  * Emergency Department visit for any reason
  * Reoperation

CONTACTS AND LOCATIONS:
Overall Officials: Jay Agarwal, MD, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (1):
- University of Utah Huntsman Cancer Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Statistics NCfDA. Opioid Epidemic: Addiction Statistics. Accessed February 16, 2024, https://drugabusestatistics.org/opioid-epidemic/
- [Background] Marcusa DP, Mann RA, Cron DC, Fillinger BR, Rzepecki AK, Kozlow JH, Momoh A, Englesbe M, Brummett C, Waljee JF. Prescription Opioid Use among Opioid-Naive Women Undergoing Immediate Breast Reconstruction. Plast Reconstr Surg. 2017 Dec;140(6):1081-1090. doi: 10.1097/PRS.0000000000003832. PMID 29176408
- [Background] Samuel AR, Fuhr L, DeGeorge BR Jr, Black J, Campbell C, Stranix JT. Prolonged Opioid Use Among Opioid-Naive Women Undergoing Breast Reconstructive Surgery. Arch Plast Surg. 2022 May 27;49(3):339-345. doi: 10.1055/s-0042-1744419. eCollection 2022 May. PMID 35832151
- [Background] (OPEN) OPEN. OPEN Prescribing Recommendations. This document was retrieved from a website with the URL: https://doi.org/10.56137/OPEN.000054
- [Background] Batdorf NJ, Lemaine V, Lovely JK, Ballman KV, Goede WJ, Martinez-Jorge J, Booth-Kowalczyk AL, Grubbs PL, Bungum LD, Saint-Cyr M. Enhanced recovery after surgery in microvascular breast reconstruction. J Plast Reconstr Aesthet Surg. 2015 Mar;68(3):395-402. doi: 10.1016/j.bjps.2014.11.014. Epub 2014 Nov 21. PMID 25488326
- [Background] Muetterties CE, Taylor JM, Kaeding DE, Morales RR, Nguyen AV, Kwan L, Tseng CY, Delong MR, Festekjian JH. Enhanced Recovery after Surgery Protocol Decreases Length of Stay and Postoperative Narcotic Use in Microvascular Breast Reconstruction. Plast Reconstr Surg Glob Open. 2023 Dec 14;11(12):e5444. doi: 10.1097/GOX.0000000000005444. eCollection 2023 Dec. PMID 38098953
- [Background] Pierzchajlo N, Zibitt M, Hinson C, Stokes JA, Neil ZD, Pierzchajlo G, Gendreau J, Buchanan PJ. Enhanced recovery after surgery pathways for deep inferior epigastric perforator flap breast reconstruction: A systematic review and meta-analysis. J Plast Reconstr Aesthet Surg. 2023 Dec;87:259-272. doi: 10.1016/j.bjps.2023.10.058. Epub 2023 Oct 15. PMID 37924717
- [Background] Temple-Oberle C, Shea-Budgell MA, Tan M, Semple JL, Schrag C, Barreto M, Blondeel P, Hamming J, Dayan J, Ljungqvist O; ERAS Society. Consensus Review of Optimal Perioperative Care in Breast Reconstruction: Enhanced Recovery after Surgery (ERAS) Society Recommendations. Plast Reconstr Surg. 2017 May;139(5):1056e-1071e. doi: 10.1097/PRS.0000000000003242. PMID 28445352
- [Background] Tedesco D, Mayo JL. Decreasing Opioid Prescriptions in Women Undergoing Mastectomy and Breast Reconstruction. Pain Manag Nurs. 2020 Aug;21(4):339-344. doi: 10.1016/j.pmn.2020.02.068. Epub 2020 Apr 10. PMID 32280011
- [Background] Melnyk M, Casey RG, Black P, Koupparis AJ. Enhanced recovery after surgery (ERAS) protocols: Time to change practice? Can Urol Assoc J. 2011 Oct;5(5):342-8. doi: 10.5489/cuaj.11002. PMID 22031616
- [Background] Kadakia NN, Rogers RL, Reed JB, Dark ER, Plake KI. Patient education interventions for prescription opioids: A systematic review. J Am Pharm Assoc (2003). 2020 Jul-Aug;60(4):e31-e42. doi: 10.1016/j.japh.2020.02.013. Epub 2020 Apr 3. PMID 32253087
- [Background] Rose KR, Christie BM, Block LM, Rao VK, Michelotti BF. Opioid Prescribing and Consumption Patterns following Outpatient Plastic Surgery Procedures. Plast Reconstr Surg. 2019 Mar;143(3):929-938. doi: 10.1097/PRS.0000000000005351. PMID 30817667
- [Background] Zhang KK, Blum KM, Chu JJ, Sharma S, Skoracki RJ, Moore AM, Janis JE, Barker JC. Reducing Opioid Overprescribing through Procedure-specific Prescribing Guidelines. Plast Reconstr Surg Glob Open. 2023 Jan 20;11(1):e4776. doi: 10.1097/GOX.0000000000004776. eCollection 2023 Jan. PMID 36699205
- [Background] Goldberg RF. The Opioid Crisis: The Surgeon's Role. Adv Surg. 2019 Sep;53:305-325. doi: 10.1016/j.yasu.2019.04.015. Epub 2019 May 17. No abstract available. PMID 31327454
- [Background] Hah JM, Bateman BT, Ratliff J, Curtin C, Sun E. Chronic Opioid Use After Surgery: Implications for Perioperative Management in the Face of the Opioid Epidemic. Anesth Analg. 2017 Nov;125(5):1733-1740. doi: 10.1213/ANE.0000000000002458. PMID 29049117
- [Background] Sun EC, Darnall BD, Baker LC, Mackey S. Incidence of and Risk Factors for Chronic Opioid Use Among Opioid-Naive Patients in the Postoperative Period. JAMA Intern Med. 2016 Sep 1;176(9):1286-93. doi: 10.1001/jamainternmed.2016.3298. PMID 27400458
- [Background] Bartels K, Mayes LM, Dingmann C, Bullard KJ, Hopfer CJ, Binswanger IA. Opioid Use and Storage Patterns by Patients after Hospital Discharge following Surgery. PLoS One. 2016 Jan 29;11(1):e0147972. doi: 10.1371/journal.pone.0147972. eCollection 2016. PMID 26824844
- [Background] Bicket MC, Long JJ, Pronovost PJ, Alexander GC, Wu CL. Prescription Opioid Analgesics Commonly Unused After Surgery: A Systematic Review. JAMA Surg. 2017 Nov 1;152(11):1066-1071. doi: 10.1001/jamasurg.2017.0831. PMID 28768328
- [Background] Howard R, Fry B, Gunaseelan V, Lee J, Waljee J, Brummett C, Campbell D Jr, Seese E, Englesbe M, Vu J. Association of Opioid Prescribing With Opioid Consumption After Surgery in Michigan. JAMA Surg. 2019 Jan 1;154(1):e184234. doi: 10.1001/jamasurg.2018.4234. Epub 2019 Jan 16. PMID 30422239
- [Background] Edwards DA, Hedrick TL, Jayaram J, Argoff C, Gulur P, Holubar SD, Gan TJ, Mythen MG, Miller TE, Shaw AD, Thacker JKM, McEvoy MD; POQI-4 Working Group. American Society for Enhanced Recovery and Perioperative Quality Initiative Joint Consensus Statement on Perioperative Management of Patients on Preoperative Opioid Therapy. Anesth Analg. 2019 Aug;129(2):553-566. doi: 10.1213/ANE.0000000000004018. PMID 30768461
- [Background] Howard R, Brown CS, Lai YL, Gunaseelan V, Brummett CM, Englesbe M, Waljee J, Bicket MC. Postoperative Opioid Prescribing and New Persistent Opioid Use: The Risk of Excessive Prescribing. Ann Surg. 2023 Jun 1;277(6):e1225-e1231. doi: 10.1097/SLA.0000000000005392. Epub 2022 Jan 21. PMID 35129474
- [Background] Waljee JF, Li L, Brummett CM, Englesbe MJ. Iatrogenic Opioid Dependence in the United States: Are Surgeons the Gatekeepers? Ann Surg. 2017 Apr;265(4):728-730. doi: 10.1097/SLA.0000000000001904. No abstract available. PMID 27429023
- [Background] Crystal DT, Cuccolo NG, Plewinski MJ, Ibrahim AMS, Sinkin JC, Lin SJ, Agag RL, Lee BT. Assessment of Opioid-Prescribing Practices in Breast Augmentation: Future Directions for Prescribing Guidelines. Ann Plast Surg. 2021 Jan;86(1):11-18. doi: 10.1097/SAP.0000000000002430. PMID 32568754
- [Background] Upp LA, Waljee JF. The Opioid Epidemic. Clin Plast Surg. 2020 Apr;47(2):181-190. doi: 10.1016/j.cps.2019.12.005. PMID 32115045
- [Background] Ghaddaf AA, Alsharef JF, Alhindi AK, Bahathiq DM, Khaldi SE, Alowaydhi HM, Alshehri MS. Influence of perioperative opioid-related patient education: A systematic review and meta-analysis. Patient Educ Couns. 2022 Sep;105(9):2824-2840. doi: 10.1016/j.pec.2022.04.016. Epub 2022 May 4. PMID 35537899
- [Background] Zorrilla-Vaca A, Mena GE, Ramirez PT, Lee BH, Sideris A, Wu CL. Effectiveness of Perioperative Opioid Educational Initiatives: A Systematic Review and Meta-Analysis. Anesth Analg. 2022 May 1;134(5):940-951. doi: 10.1213/ANE.0000000000005634. PMID 34125081
- [Background] Health NIo. Plain Language at NIH. Accessed February 15, 2024, https://www.nih.gov/institutes-nih/nih-office-director/office-communications-public-liaison/clear-communication/plain-language
- [Background] Amtmann D, Cook KF, Jensen MP, Chen WH, Choi S, Revicki D, Cella D, Rothrock N, Keefe F, Callahan L, Lai JS. Development of a PROMIS item bank to measure pain interference. Pain. 2010 Jul;150(1):173-182. doi: 10.1016/j.pain.2010.04.025. PMID 20554116
- [Background] Askew RL, Cook KF, Revicki DA, Cella D, Amtmann D. Evidence from diverse clinical populations supported clinical validity of PROMIS pain interference and pain behavior. J Clin Epidemiol. 2016 May;73:103-11. doi: 10.1016/j.jclinepi.2015.08.035. Epub 2016 Feb 27. PMID 26931296
- [Background] Revicki DA, Chen WH, Harnam N, Cook KF, Amtmann D, Callahan LF, Jensen MP, Keefe FJ. Development and psychometric analysis of the PROMIS pain behavior item bank. Pain. 2009 Nov;146(1-2):158-69. doi: 10.1016/j.pain.2009.07.029. Epub 2009 Aug 15. PMID 19683873
- [Background] Stone AA, Broderick JE, Junghaenel DU, Schneider S, Schwartz JE. PROMIS fatigue, pain intensity, pain interference, pain behavior, physical function, depression, anxiety, and anger scales demonstrate ecological validity. J Clin Epidemiol. 2016 Jun;74:194-206. doi: 10.1016/j.jclinepi.2015.08.029. Epub 2015 Nov 25. PMID 26628334
- [Background] HealthMeasures. Intro to PROMIS®. Accessed February 16, 2024, https://www.healthmeasures.net/explore-measurement-systems/promis/intro-to-promis
- [Background] BREAST-Q | BREAST CANCER. Accessed February 16, 2024, https://qportfolio.org/breast-q/breast-cancer/
- [Background] Cano SJ, Klassen AF, Scott AM, Cordeiro PG, Pusic AL. The BREAST-Q: further validation in independent clinical samples. Plast Reconstr Surg. 2012 Feb;129(2):293-302. doi: 10.1097/PRS.0b013e31823aec6b. PMID 22286412
- [Background] Fuzesi S, Cano SJ, Klassen AF, Atisha D, Pusic AL. Validation of the electronic version of the BREAST-Q in the army of women study. Breast. 2017 Jun;33:44-49. doi: 10.1016/j.breast.2017.02.015. Epub 2017 Mar 7. PMID 28279888
- [Background] Kaur MN, Chan S, Bordeleau L, Zhong T, Tsangaris E, Pusic AL, Cano SJ, Klassen AF. Re-examining content validity of the BREAST-Q more than a decade later to determine relevance and comprehensiveness. J Patient Rep Outcomes. 2023 Apr 6;7(1):37. doi: 10.1186/s41687-023-00558-y. PMID 37022647
- [Background] Maheu AR, Hohmann AL, Cozzarelli NF, Khan IA, Hozack WJ, Ilyas AM, Lonner JH. The Efficacy of Preoperative Video-Based Opioid Counseling on Postoperative Opioid Consumption After Total Knee Arthroplasty: A Prospective Randomized Controlled Trial. J Arthroplasty. 2024 Aug;39(8S1):S143-S147. doi: 10.1016/j.arth.2024.02.027. Epub 2024 Feb 24. PMID 38403081
- [Background] Marquez JL, Chow J, Moss W, Luo J, Eddington D, Agarwal JP, Kwok AC. Outpatient Prescription Opioid Use following Discharge after Deep Inferior Epigastric Perforator Breast Reconstruction with and without an Educational Intervention. J Reconstr Microsurg. 2024 Nov;40(9):688-693. doi: 10.1055/a-2283-4775. Epub 2024 Mar 7. PMID 38452802
- [Background] Egan KG, De Souza M, Muenks E, Nazir N, Korentager R. Predictors of Opioid Consumption in Immediate, Implant-Based Breast Reconstruction. Plast Reconstr Surg. 2020 Oct;146(4):734-741. doi: 10.1097/PRS.0000000000007150. PMID 32969995